CLINICAL TRIAL: NCT01893320
Title: A Phase I/II Study of Vosaroxin and Decitabine in Older Patients With Acute Myeloid Leukemia and High-risk Myelodysplastic Syndrome
Brief Title: Study of Vosaroxin and Decitabine in Older Patients With Acute Myeloid Leukemia and High-risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0099; NCI-2013-01665 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia; AML; High-risk Myelodysplastic Syndrome; MDS; Chronic Myelomonocytic Leukemia; CMM; Maximum tolerated dose; MTD; Vosaroxin; Decitabine; Dacogen
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — vosaroxin; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vosaroxin + Decitabine (Experimental): The first 6 patients on study (first cohort) receive 1 or 2 induction cycles of therapy according to the following starting schedule: Vosaroxin administered intravenously on days 1 and 4 at a dose of 90 mg/m2 in the first cycle (induction 1) for a total dose of 180 mg/m2/cycle in combination with Decitabine at a dose of 20 mg/m2 intravenously daily for 5 consecutive days (Days 1 to 5).
  Following the phase I portion, patients in phase II receive the following induction:
  1. Vosaroxin intravenously on days 1 and 4 at a dose of 70 mg/m2 for a total dose of 140 mg/m2/cycle (days 1 and 4), or the final induction dose (MTD) determined in phase I.
  2. Decitabine intravenously at a dose of 20 mg/m2 for 5 consecutive days (days 1 to 5), or the final induction dose (MTD) determined in phase I.
  Interventions: Drug: Vosaroxin; Drug: Decitabine

INTERVENTIONS:
Drug: Vosaroxin — Phase I Starting Dose: 90 mg/m2 by vein on Days 1 and 4 of each cycle.
  Phase II Starting Dose: 70 mg/m2 by vein on Days 1 and 4 of each cycle, or maximum tolerated dose from Phase I.
Drug: Decitabine — Phase I and II: 20 mg/m2 by vein daily for 5 consecutive days (Days 1 to 5).
  Other Names: Dacogen

SUMMARY:
The goal of this clinical research study is to learn if the combination of vosaroxin and decitabine can help to control AML or MDS. The safety of these drugs will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 4 groups of up to 6 participants will be enrolled in the Phase I portion of the study, and up to 60 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of vosaroxin you receive will depend on when you joined this study. The first group of participants will receive the highest dose level of vosaroxin. If no intolerable side effects are seen, the study will move on to Phase II. If intolerable side effects are seen, each new group will receive a lower dose of vosaroxin than the group before it until the most tolerable dose is found.

If you are enrolled in the Phase II portion, you will receive vosaroxin at the highest dose that was tolerated in the Phase I portion.

All participants will receive the same dose level of decitabine.

Study Drug Administration:

You will receive the study drugs in cycles. The study cycles will be 4-12 weeks long, depending on if/how the disease responds to the treatment, how your bone marrow reacts to treatment, and what the doctor thinks is in your best interest.

On Days 1-5 of each study cycle, you will receive decitabine by vein over about 1 hour. On Days 1 and 4 of each cycle, you will also receive vosaroxin by vein over 8-10 minutes, before you receive decitabine. Depending on how the disease responds to the study drugs, the number of days you receive the study drug may change. Your doctor will discuss this with you.

The first 2 cycles are called Induction Cycles. All cycles after that are called Consolidation Cycles. All participants will receive Induction Cycle 1. If the study doctor thinks it is needed, you will also receive Induction Cycle 2. If after that the study doctor thinks it is in your best interest, you will receive up to 5 Consolidation Cycles of treatment.

Study Visits:

On Day 1 of each cycle, you will have a physical exam.

Every week, blood (about 1 tablespoon) will be drawn for routine tests. If at any point you appear to have a response to the study drugs, this blood will then be drawn every 1-2 weeks while you are still receiving the study drugs. If your doctor thinks it is needed, more blood may need to be drawn.

On Day 21 of Cycle 1 (+/- 7 days), then every 4 weeks after that, you will have a bone marrow aspiration and/or biopsy to check the status of the disease. If the doctor thinks it is needed, these may be done more or less often, depending on your response to the study drugs.

Length of Study:

You may receive the study drugs for up to 7 cycles. You will be taken off study if the disease gets worse, intolerable side effects occur, or if the study doctor thinks it is in your best interest.

Your participation in the study will be over after the follow-up period.

End-of-Study Visit:

If you are taken off study or if you leave the study early, you will have an end-of-study visit. At this visit:

Blood (about 2-3 teaspoons) will be drawn for routine tests. If the study doctor thinks it is needed, you will have a bone marrow aspiration.

You will then be contacted during a study visit or called and asked about any side effects you may be having 30 days after the end-of-study visit. This call will last about 5 minutes.

Follow-up:

If you do not leave the study early, you will have follow-up visits and calls for up to 5 years after you stop receiving the study drugs.

Every 4-8 weeks, blood (about 1 tablespoon) will be drawn for routine tests. If you cannot return to the clinic, you may have blood drawn at a clinic close to your home.

Every 3-6 months, you will be contacted during a clinic visit and asked how you are doing. If you cannot make it to the clinic for this visit, you will be called. The phone call should last about 5 minutes.

This is an investigational study. Vosaroxin is not FDA approved or commercially available. It is currently being used for research purposes only. Decitabine has been approved by the FDA for the treatment of MDS, which is a precursor of AML, but has not been approved for the treatment of AML. The use of these drugs in combination is investigational. The study doctor can explain how the drugs are designed to work.

Up to 84 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated AML (>/= 20% blasts). Patients with high-risk MDS (defined as having >/= 10% blasts in the bone marrow) or patients with Chronic Myelomonocytic Leukemia (CMML) (having >/= 10% blasts in the bone marrow) may also be eligible after discussion with Principal Investigator (PI). Prior therapy with hydroxyurea, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is allowed, however prior therapy with chemotherapy agents for the disease under study is not allowed. Patients may have received one dose of cytarabine (up to 2 g/m2) administered at presentation for control of hyperleucocytosis. For patients with prior MDS or CMML who transformed to AML, therapy received for MDS is not considered as prior therapy for AML.
2. Age >/= 60 years and not candidates for conventional cytotoxic chemotherapy or refuse it; OR patients below the age of 60 years who are considered unfit and/or unable to tolerate standard chemotherapy at the discretion of the treating physician or the principal investigator. "
3. Eastern Cooperative Oncology Group performance status </= 2.
4. Adequate hepatic (serum total bilirubin </= 1.5 x upper limit normal (ULN), alanine aminotransferase and/or aspartate transaminase </= 2.5 x ULN) and renal function (creatinine </= 2.0 mg/dL).
5. Left ventricular ejection fraction (LVEF) at least 40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
6. Patients must be willing and able to review, understand, and provide written consent before starting therapy.
7. Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum pregnancy test within 14 days before the start of the treatment. Women of childbearing potential may have a urine pregnancy test, instead of a serum pregnancy test. If either the serum or urine pregnancy test is equivocally negative the patient will be eligible for the protocol. Women of childbearing potential must agree to use an adequate method of contraception during the study until 30 days after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 30 days after the last treatment.

Exclusion Criteria:

1. New York Heart Association class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as active angina pectoris, clinically significant cardiac arrhythmia that requires therapy in the opinion of the treating physician or PI, uncontrolled hypertension (blood pressure > 160 systolic and > 110 diastolic not responsive to antihypertensive medication), uncontrolled diabetes mellitus in the opinion of the treating physician or PI, or uncontrolled congestive heart failure in the opinion of the treating physician or PI.
2. Myocardial infarction in the previous 12 weeks (from the start of treatment).
3. Active and uncontrolled disease/infection as judged by the treating physician
4. Pregnant or breastfeeding
5. Known Human Immunodeficiency Virus seropositivity
6. Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator or medical monitor
7. Acute promyelocytic leukemia (APL).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-07-18 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Daver N, Kantarjian H, Garcia-Manero G, Jabbour E, Borthakur G, Brandt M, Pierce S, Vaughan K, Ning J, Nogueras Gonzalez GM, Patel K, Jorgensen J, Pemmaraju N, Kadia T, Konopleva M, Andreeff M, DiNardo C, Cortes J, Ward R, Craig A, Ravandi F. Vosaroxin in combination with decitabine in newly diagnosed older patients with acute myeloid leukemia or high-risk myelodysplastic syndrome. Haematologica. 2017 Oct;102(10):1709-1717. doi: 10.3324/haematol.2017.168732. Epub 2017 Jul 20. PMID 28729302
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2013 to June 2016
Groups:
- Phase I MTD Vosaroxin: The first 7 patients on study (first cohort) receive 1 or 2 induction cycles of therapy according to the following starting schedule: Vosaroxin administered intravenously on days 1 and 4 at a dose of 90 mg/m2 in the first cycle (induction 1) for a total dose of 180 mg/m2/cycle in combination with Decitabine at a dose of 20 mg/m2 intravenously daily for 5 consecutive days (Days 1 to 5).
- Vosaroxin + Decitabine: The first 7 patients on study (first cohort) receive 1 or 2 induction cycles of therapy according to the following starting schedule: Vosaroxin administered intravenously on days 1 and 4 at a dose of 90 mg/m2 in the first cycle (induction 1) for a total dose of 180 mg/m2/cycle in combination with Decitabine at a dose of 20 mg/m2 intravenously daily for 5 consecutive days (Days 1 to 5).
  Following the phase I portion, patients in phase II receive the following induction:
  1. Vosaroxin intravenously on days 1 and 4 at a dose of 70 mg/m2 for a total dose of 140 mg/m2/cycle (days 1 and 4), or the final induction dose (MTD) determined in phase I.
  2. Decitabine intravenously at a dose of 20 mg/m2 for 5 consecutive days (days 1 to 5), or the final induction dose (MTD) determined in phase I.
  Vosaroxin: Phase I Starting Dose: 90 mg/m2 by vein on Days 1 and 4 of each cycle.
  Phase II Starting Dose: 70 mg/m2 by vein on Days 1 and 4 of each cycle, or maximum tolerated dose from Phase I.
  Decitabine: Phase I and II: 20 mg/m2 by vein daily for 5 consecutive days (Days 1 to 5).
Period: Overall Study
Arm/Group | Phase I MTD Vosaroxin | Vosaroxin + Decitabine
Started | 7 | 59
Completed | 7 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I MTD Vosaroxin | Vosaroxin + Decitabine | Total
Number analyzed (Participants) | 7 | 59 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 9 | 11
  >=65 years | 5 | 50 | 55
Age, Continuous [Median (Full Range); unit: years] | 69 [41 to 75] | 69 [60 to 78] | 69 [41 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 24 | 24
  Male | 7 | 35 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 7 | 49 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 59 | 66

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Vosaroxin in Combination With Decitabine
Description: Maximum tolerated dose (MTD) defined as highest daily oral dose evaluated at which <33% of patients experience a dose limiting toxicity (DLT). A non-hematologic dose-limiting toxicity (DLT) defined as a clinically significant grade 3 or 4 adverse event or abnormal laboratory value (according to CTCAE criteria) assessed by treating physician as related to study drug (and unrelated to disease progression, intercurrent illness, or concomitant medications) occurring during the first 28 days on study. A hematologic DLT defined as severe myelosuppression with a hypoplastic marrow with less than 5% cellularity and no evidence of leukemia 42 days from start of therapy. This will define severe and delayed myelosuppression not related to persistent leukemia and likely related to treatment.
Time Frame: 21 days
Measure: Number; unit: Mg/m^2
Arm/Group | Phase I MTD Vosaroxin
Number analyzed (Participants) | 7
Mg/m^2 | 70

2. Secondary Outcome: Participants With a Response
Description: A Response is defined as: Complete response (CR) + Complete response without platelet recovery (CRp) + CR with insufficient hematological recovery (platelets or neutrophils (CRi). CR is Neutrophil count 2: 1.0 x 10^9/L, platelet count 2: 100 x 10^9/L and bone marrow aspirate and biopsy: S5% blasts. CRp is same as CR but with Platelets < 100 x 10^/L. CRi is same as CR but platelets < 100 x 10(/L or neutrophils < 1 x 10^9.
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I MTD Vosaroxin | Vosaroxin + Decitabine
Number analyzed (Participants) | 7 | 59
Participants | 7 | 42

ADVERSE EVENTS:
Time Frame: Up to 2 years 11 months
Groups:
- Vasoroxin + Decitabine: The first 7 patients on study (first cohort) receive 1 or 2 induction cycles of therapy according to the following starting schedule: Vosaroxin administered intravenously on days 1 and 4 at a dose of 90 mg/m2 in the first cycle (induction 1) for a total dose of 180 mg/m2/cycle in combination with Decitabine at a dose of 20 mg/m2 intravenously daily for 5 consecutive days (Days 1 to 5).
  Following the phase I portion, patients in phase II receive the following induction:
  1. Vosaroxin intravenously on days 1 and 4 at a dose of 70 mg/m2 for a total dose of 140 mg/m2/cycle (days 1 and 4), or the final induction dose (MTD) determined in phase I.
  2. Decitabine intravenously at a dose of 20 mg/m2 for 5 consecutive days (days 1 to 5), or the final induction dose (MTD) determined in phase I.
  Vosaroxin: Phase I Starting Dose: 90 mg/m2 by vein on Days 1 and 4 of each cycle.
  Phase II Starting Dose: 70 mg/m2 by vein on Days 1 and 4 of each cycle, or maximum tolerated dose from Phase I.
  Decitabine: Phase I and II: 20 mg/m2 by vein daily for 5 consecutive days (Days 1 to 5).
Arm/Group | Phase I MTD Vosaroxin | Vasoroxin + Decitabine
All-Cause Mortality (participants affected / at risk) | 0/7 | 7/59
Serious Adverse Events (participants affected / at risk) | 6/7 | 48/59
Other Adverse Events (participants affected / at risk) | 2/7 | 19/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I MTD Vosaroxin (N=7) | Vasoroxin + Decitabine (N=59)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 2 (2)
Bone Infection (Infections and infestations) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Catheter Related Infection (Infections and infestations) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Edema Face (General disorders) | 0 (0) | 1 (1)
Enterocolitis Infection (Infections and infestations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (8) | 18 (23)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized Weakness (General disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 8 (10)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2) | 13 (17)
Mucositis Oral (Gastrointestinal disorders) | 2 (2) | 4 (4)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 11 (12)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I MTD Vosaroxin (N=7) | Vasoroxin + Decitabine (N=59)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increase (Investigations) | 0 (0) | 1 (1)
Blood Bilirubin Increase (Investigations) | 1 (1) | 2 (2)
Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Dysartharia (Nervous system disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Hallucinations (Nervous system disorders) | 0 (0) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Hoarsness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT01893320/Prot_SAP_000.pdf